CLINICAL TRIAL: NCT04495868
Title: Bacteriostatic Normal Saline Versus Lidocaine for Intradermal Anesthesia During Lumbar Medial Branch Block
Brief Title: Bacteriostatic Normal Saline Versus Lidocaine for Intradermal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brian Bobzien, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00000428
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain
Keywords: Local anesthetic
MeSH Terms: conditions — Chronic Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bacteriostatic Normal Saline then 1% Lidocaine (Experimental): Participants undergoing a lumbar medial branch block who are randomized to receive an intradermal administration of bacteriostatic normal saline followed by an intradermal administration of 1% lidocaine.
  Interventions: Drug: Bacteriostatic Normal Saline; Drug: 1% Lidocaine
- 1% Lidocaine then Bacteriostatic Normal Saline (Active Comparator): Participants undergoing a lumbar medial branch block who are randomized to receive an intradermal administration of 1% lidocaine followed by an intradermal administration of bacteriostatic normal saline.
  Interventions: Drug: Bacteriostatic Normal Saline; Drug: 1% Lidocaine

INTERVENTIONS:
Drug: Bacteriostatic Normal Saline — A skin wheal will be made with bacteriostatic normal saline (BNS). BNS contains 0.9% benzyl alcohol and benzyl alcohol is an opium alkaloid that is sometimes added to physiologic normal saline for its bacteriostatic properties. The skin wheal will be created by injecting the medication intra-dermally with a 26 gauge needle.
Drug: 1% Lidocaine — A skin wheal will be made with 1% lidocaine. The skin wheal will be created by injecting the medication intra-dermally with a 26 gauge needle.

SUMMARY:
The purpose of this study is to determine if creation of a skin wheel with bacteriostatic normal saline, which includes 0.9% benzyl alcohol, is less painful and provides a similar level of anesthesia compared to 1% lidocaine. Participants will receive both types of anesthesia, in random order.

DETAILED DESCRIPTION:
Most chronic pain procedures or injections utilize medications (e.g. local anesthetics) to numb the skin in an effort to reduce procedure-related pain; however, they can also be a significant cause of pain leading the patient to abort the procedure. Studies have looked at alternative medications and techniques that lessen the pain but still provide similar levels of anesthesia ("numbing"). One such alternative medication is normal saline that includes benzyl alcohol. Studies researching this specific medication have usually examined procedural pain related to drawing blood or placing an intravenous (IV) catheter but not for chronic pain related procedures.

This is a single site randomized double-blinded clinical trial that will compare the standard of care (1% lidocaine) with bacteriostatic normal saline (saline with benzyl alcohol) administered as a skin wheal during a diagnostic procedure in patients with chronic low back pain. The order of administration of the medication will be randomized and the medication will be blinded to both the subject and the investigator performing the procedure. Skin wheals will be created with each medication, and the subject's level of pain will be assessed after each one to measure how painful the creation of the skin wheal was. Then, a spinal needle for the diagnostic procedure will be placed through the skin wheal and the subject's level of pain will be assessed after each one to measure the level of anesthesia (or numbing) that each one provides. The objectives of this study are to determine if administration of bacteriostatic normal saline causes less discomfort than 1% lidocaine and provides a similar level of anesthesia/numbing for the procedure.

The study will take place at the Grady Pain clinic and participants will be identified from patients that are scheduled to undergo a specific low back procedure - diagnostic lumbar medial branch block. This research study will help identify potential alternatives to the standard of care for numbing of skin during chronic pain procedures that may reduce procedure-related pain and discomfort thus making the procedure more tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an initial lumbar medial branch block

Exclusion Criteria:

* Allergy to local anesthetics
* Fibromyalgia
* Inability to provide informed consent in English
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Bobzien, MD, Principal Investigator — Emory University
Locations (1):
- Grady Pain Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial will be available for sharing, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available for sharing beginning immediately upon publication and ending 36 months following article publication.
Access Criteria: Data will be available for sharing with researchers who provide a methodologically sound proposal, in order to achieve the aims in the approved proposal. Proposals should be directed to bbobzie@emory.edu. A link will be provided to the researcher for download of the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bacteriostatic Normal Saline Then 1% Lidocaine | 1% Lidocaine Then Bacteriostatic Normal Saline
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bacteriostatic Normal Saline Then 1% Lidocaine | 1% Lidocaine Then Bacteriostatic Normal Saline | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 20 | 34
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 6 | 2 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40
Numerical Pain Rating Scale (NPRS) Score of Back Pain [Median (Inter-Quartile Range); unit: units on a scale] — The NPRS is an 11-point, self-rated pain scale where participants rate the level of their chronic axial low back pain from 0 (no pain) to 10 (worst pain imaginable).
  units on a scale | 8 [7 to 8] | 8 [6 to 8] | 8 [6 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Needle Placement Pain Score
Description: Participants rated their pain level from the insertion of the needle for the lumbar medial branch block using the skin wheal created with each anesthetic. Pain is rated on a scale from 0 to 10, where 0 = no pain and 10 = worst pain.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Bacteriostatic Normal Saline: Participants undergoing a lumbar medial branch block receiving an intradermal administration of bacteriostatic normal saline.
- 1% Lidocaine: Participants undergoing a lumbar medial branch block receiving an intradermal administration of 1% lidocaine.
Arm/Group | Bacteriostatic Normal Saline | 1% Lidocaine
Number analyzed (Participants) | 40 | 40
units on a scale | 0 [0 to 1] | 0 [0 to 0]

2. Secondary Outcome: Skin Wheal Pain Score
Description: Participants rated their pain level from the creation of the skin wheal using each anesthetic on a scale from 0 to 10, where 0 = no pain and 10 = worst pain.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bacteriostatic Normal Saline | 1% Lidocaine
Number analyzed (Participants) | 40 | 40
units on a scale | 5 [2 to 7] | 6 [4 to 9]

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected during the lumbar medial branch block procedure (Day 1 of study).
Arm/Group | Bacteriostatic Normal Saline | 1% Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT04495868/Prot_SAP_000.pdf